CLINICAL TRIAL: NCT03807011
Title: The Effects of Remifentanil and Fentanyl on Emergence Agitation in Pediatric Strabismus Surgery
Brief Title: Emergence Agitation in Pediatric Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Eun Kyung Choi, Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YUMC 2017-04-071
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Emergence Agitation
Keywords: Emergence Agitation; fentanyl; remifentanil; children
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fentanyl (Active Comparator): A bolus dose of fentanyl 2 μg/kg was administered intravenously at anesthetic induction
  Interventions: Drug: fentanyl group
- remifentanil (Active Comparator): Remifentanil was continuously infused at a rate of 0.2 μg/kg/min from anesthetic induction to the end of surgery
  Interventions: Drug: remifentanil group

INTERVENTIONS:
Drug: fentanyl group — fentanyl 2 μg/kg
  Arms: fentanyl
Drug: remifentanil group — remifentanil 0.2 μg/kg/min
  Arms: remifentanil

SUMMARY:
This study was performed to assess the effects of continuous remifentanil infusion and single bolus administration of fentanyl on the incidence of emergence agitation in pediatrics undergoing strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective subumbilical surgery,
* physical status was American Society of Anesthesiologists (ASA) class 1 or 2

Exclusion Criteria:

* history of airway problem,
* upper respiratory tract infection within 2 weeks,
* developmental delay,
* neurological or psychological disease,
* history of allergy to the drugs in our protocol were excluded in this study.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative agitation | 5 minutes in the recovery room
  0=none; 1=occur
incidence of postoperative agitation | 30 minutes in the recovery room
  0=none; 1=occur
severity of postoperative agitation | 5 minutes in the recovery room
  Four-point agitation scale (0=calm; 1=not calm but could easily become calmed; 3=not easily calmed, moderately agitated and restless; 4=combative, excited, or disoriented)
severity of postoperative agitation | 30 minutes in the recovery room
  Four-point agitation scale (0=calm; 1=not calm but could easily become calmed; 3=not easily calmed, moderately agitated and restless; 4=combative, excited, or disoriented)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Eun kyung Choi, Daegu, Korea (the Republic Of)
  - Yeungnam University Hospital, Daegu, Nam-gu, Daegu